CLINICAL TRIAL: NCT03332979
Title: Experiencing Loss and Planning Ahead Study (ELPAS): Caring for a Relative or Friend With Dementia
Brief Title: Experiencing Loss and Planning Ahead Study
Acronym: ELPAS
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Alzheimer's Society (Other)
Responsible Party: Sponsor
Other Study IDs: 17/0477
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Grief
Keywords: pre-death grief; palliative care; dementia; caregiver; preparation for end of life
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The course of dementia over many years, gradual losses and uncertain life expectancy can lead to grief amongst family and friend carers. This study aims to examine the relationship between carers' feelings of grief before the death of a person with dementia and how well carers are prepared for that death. The study involves completing questionnaires with 150 carers of people with dementia (at home or in a care home). Twenty of these carers will be purposively selected to complete additional semi-structured questions to further explore the research questions. The questionnaires will examine whether being prepared for end of life is linked to having lower levels of grief. Preparation will be measured by important factors shown in research including: knowledge of dementia progression; knowledge of the person with dementia's end of life preferences; communication with healthcare professionals; family support; and having a Power of Attorney or advance directives. The study is part of a larger study that will also involve surveys with service providers and developing a resource for carers. The study will provide important insights into how we can better support grieving carers and help them plan and prepare for end of life care.

DETAILED DESCRIPTION:
Grief is often felt before the death of a friend or relative with dementia. Grief before the death can be triggered by losses associated with dementia causing carers to experience sorrow, anger, yearning and acceptance that can wax and wane from diagnosis to the end of life. It occurs due to the lengthy and uncertain disease trajectory; compromised communication between the person with dementia and family and friends; and changes in relationship quality and carer freedom. Between 47-71% of family and friends of people with dementia (referred here as 'carers') experience grief before the death and 20% experience complicated grief after the death. Higher grief prior to death is associated with complicated grief after death, so emotional support during care rather than solely after the death may be beneficial.

Preparation for end of life has medical, psychosocial, spiritual and practical components, including having a family member or healthcare professional to help make decisions, knowing what to expect about the terminal condition and having finances in place. Good communication with healthcare providers to discuss prognosis, treatments, cultural, spiritual and practical issues; and dealing with family conflict is critical. Preparation for end of life is associated with a lower likelihood of complicated grief in bereavement but has not been explored in the context of grief before the death. Preparation for end of life is influenced by socioeconomic factors associated with health literacy. In the UK a third of older adults have difficulty interpreting basic health information. Despite the potential benefits of end of life discussions with carers, there are many barriers to such discussions. Carers struggle to formalise in writing future wishes on behalf of the person with dementia and professionals tend to be reluctant to initiate end of life discussions. Family conflict can deter end of life decision making. Factors reflecting preparation for end of life are potentially modifiable suggesting that improving preparation could reduce grief before the death.

This study aims to examine the relationship between family and friend carers' feelings of grief before the death of a person with dementia and how well carers are prepared for that death. The hypothesis that will be tested is that modifiable factors indicating preparation for end of life are associated with lower grief before the death in carers of people with dementia. The modifiable factors reflecting preparation for end of life include: carers' having a good knowledge of dementia progression; high health literacy; a lasting (enduring) Power of Attorney; knowing the end of life wishes of the person with dementia; being satisfied with support from their social network.

Knowing which modifiable factors reflecting preparation for end of life are most closely associated with grief before the death will inform the development of a resource for carers with the potential to reduce carer distress during the lifetime of the person with dementia, bringing benefits for the person with dementia as well as their carer. It will enable discussions to ensure care at the end of life is planned and in accordance with the person's wishes; and may reduce the prevalence of complicated grief after the death of the person with dementia.

Secondary objectives are to: examine the prevalence and severity of grief before the death in carers of people with dementia; identify which modifiable factors reflecting preparation for end of life are most strongly related to grief before the death; examine the extent to which carers feel prepared for the future and end-of-life care for their relative with dementia; explore whether carers recognize grief during caring and what supports they think would be helpful; identify unmet needs for information about end of life symptoms and emotional support for carers; and explore how carers experience and cope with changes in grief over time.

This is a cross-sectional study using mixed methods. One hundred and fifty carers of people with a diagnosis of dementia will be recruited to take part in the study. They will take part in a quantitative interview with a range of questionnaires. Participants will be recruited through community and healthcare services and via the Join Dementia Research Register in the United Kingdom. Eligible carers will be sent invitations to participate. Flyers in these services or presentations at family meetings of these services are other potential avenues for recruitment. Participants will provide written consent prior to the interview.

A sub-sample of carers will be asked whether they would also like to take part in an additional qualitative semi-structured interview to enable more in-depth exploration of some of the secondary objectives. The interview will explore the dynamic and changing nature of grief over time, how carers identify with the concept of grief and whether they consider they are going through a grief experience. It will also examine what supports they have found helpful and what they perceive to be unmet information and support needs and possible programs/resources that might address these needs. Qualitative interviews will be audio-recorded with permission from the participant on an encrypted digital recorder and then transcribed verbatim by the research team. Participants will be purposively selected to take part in these interviews to provide a mix of responses representing male and female participants, adult child and spouse participants, different ethnicity as well as carers of people at different severity of dementia. We will aim to interview carers until saturation of data is reached. We envisage this will be between 15-20 carers. Once we have achieved saturation we will cease inviting carers to take part in this component of the study.

For the quantitative analysis, multivariable regression analysis will be used to explore the impact of the five modifiable factors reflecting preparation for end of life on the primary outcome of pre-death grief. We will control for potential confounding variables including: dementia severity, relationship type (spouse/partner, a child or another relationship), gender, care home status (whether or not the person with dementia is living at home or in a care home), and religiosity. There are ten potential co-variates to be included in the model. A sample of 15 participants per co-variate is preferable while ten may be sufficient. We will aim to recruit 150 participants for an adequately powered analysis.

For the qualitative analysis audio-recording will be transcribed verbatim and entered into NVivo qualitative software package (QSR International) to support data coding. Data will be thematically analysed by coding chunks of text and grouping these codes into themes and sub-themes that address the study objectives. Two researchers will independently code and analyse each interview independently and then compare codes and themes to ensure rigour in analysis. Discrepancies will be discussed until consensus on themes is reached. Interviews will be coded as collected to enable subsequent interviews to draw on and explore themes arising. While we aim to recruit carers from a mix of categories (gender, relationship type and dementia severity) we will not be able to make comparisons between groups because of the small numbers representing each group (eg there may be only one male son caring for someone with mild dementia). The themes identified will help to draw out individual experiences in relation to carer grief and access to supports to supplement and expand the quantitative data.

ELIGIBILITY:
Inclusion Criteria:

* Carers of people with dementia providing practical, social, emotional or supervisory support to a friend or family member. This will include carers of people with dementia living at home or in a care home. Carers will be 18 years of age or over and living in England. The person they care for will have received a formal diagnosis of any dementia related disease.

Exclusion Criteria:

* Carers who are not able to communicate in English or who do not have capacity to provide informed written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample. Carers will be recruited via a range of services (memory services/clinics, care homes, Admiral Nurses [specialist dementia nurses] and branches of the Alzheimer's Society). Recruitment will also occur through the Join Dementia Research website which is an online register where people living in the United Kingdom can express an interest in participating in dementia research and be invited to take part in studies based on matched eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten J Moore, PhD, Principal Investigator — University College, London
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Almack K, Cox K, Moghaddam N, Pollock K, Seymour J. After you: conversations between patients and healthcare professionals in planning for end of life care. BMC Palliat Care. 2012 Sep 17;11:15. doi: 10.1186/1472-684X-11-15. PMID 22985010
- [Background] Annear MJ, Toye CM, Eccleston CE, McInerney FJ, Elliott KE, Tranter BK, Hartley T, Robinson AL. Dementia Knowledge Assessment Scale: Development and Preliminary Psychometric Properties. J Am Geriatr Soc. 2015 Nov;63(11):2375-81. doi: 10.1111/jgs.13707. Epub 2015 Oct 27. PMID 26503020
- [Background] Barry LC, Kasl SV, Prigerson HG. Psychiatric disorders among bereaved persons: the role of perceived circumstances of death and preparedness for death. Am J Geriatr Psychiatry. 2002 Jul-Aug;10(4):447-57. PMID 12095904
- [Background] Bostock S, Steptoe A. Association between low functional health literacy and mortality in older adults: longitudinal cohort study. BMJ. 2012 Mar 15;344:e1602. doi: 10.1136/bmj.e1602. PMID 22422872
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qualitative Research in Psychology 3(2): 77-101, 2006.
- [Background] Chan D, Livingston G, Jones L, Sampson EL. Grief reactions in dementia carers: a systematic review. Int J Geriatr Psychiatry. 2013 Jan;28(1):1-17. doi: 10.1002/gps.3795. Epub 2012 Mar 8. PMID 22407743
- [Background] Dening KH, Jones L, Sampson EL. Preferences for end-of-life care: a nominal group study of people with dementia and their family carers. Palliat Med. 2013 May;27(5):409-17. doi: 10.1177/0269216312464094. Epub 2012 Nov 5. PMID 23128905
- [Background] Hebert RS, Dang Q, Schulz R. Preparedness for the death of a loved one and mental health in bereaved caregivers of patients with dementia: findings from the REACH study. J Palliat Med. 2006 Jun;9(3):683-93. doi: 10.1089/jpm.2006.9.683. PMID 16752974
- [Background] Hebert RS, Prigerson HG, Schulz R, Arnold RM. Preparing caregivers for the death of a loved one: a theoretical framework and suggestions for future research. J Palliat Med. 2006 Oct;9(5):1164-71. doi: 10.1089/jpm.2006.9.1164. PMID 17040154
- [Background] Hebert RS, Schulz R, Copeland V, Arnold RM. What questions do family caregivers want to discuss with health care providers in order to prepare for the death of a loved one? An ethnographic study of caregivers of patients at end of life. J Palliat Med. 2008 Apr;11(3):476-83. doi: 10.1089/jpm.2007.0165. PMID 18363491
- [Background] Hirschman KB, Kapo JM, Karlawish JH. Identifying the factors that facilitate or hinder advance planning by persons with dementia. Alzheimer Dis Assoc Disord. 2008 Jul-Sep;22(3):293-8. doi: 10.1097/WAD.0b013e318169d669. PMID 18580595
- [Background] Lindauer A, Harvath TA. Pre-death grief in the context of dementia caregiving: a concept analysis. J Adv Nurs. 2014 Oct;70(10):2196-207. doi: 10.1111/jan.12411. Epub 2014 Apr 7. PMID 24702153
- [Background] Marwit SJ, Meuser TM. Development of a short form inventory to assess grief in caregivers of dementia patients. Death Stud. 2005 Apr;29(3):191-205. doi: 10.1080/07481180590916335. PMID 15816111
- [Background] Osborne RH, Batterham RW, Elsworth GR, Hawkins M, Buchbinder R. The grounded psychometric development and initial validation of the Health Literacy Questionnaire (HLQ). BMC Public Health. 2013 Jul 16;13:658. doi: 10.1186/1471-2458-13-658. PMID 23855504
- [Background] Petty NJ, Thomson OP, Stew G. Ready for a paradigm shift? Part 2: introducing qualitative research methodologies and methods. Man Ther. 2012 Oct;17(5):378-84. doi: 10.1016/j.math.2012.03.004. Epub 2012 Apr 3. PMID 22480949
- [Background] Romero MM, Ott CH, Kelber ST. Predictors of grief in bereaved family caregivers of person's with Alzheimer's disease: a prospective study. Death Stud. 2014 Jul-Dec;38(6-10):395-403. doi: 10.1080/07481187.2013.809031. Epub 2013 Oct 18. PMID 24666146
- [Background] Sampson EL, Jones L, Thune-Boyle IC, Kukkastenvehmas R, King M, Leurent B, Tookman A, Blanchard MR. Palliative assessment and advance care planning in severe dementia: an exploratory randomized controlled trial of a complex intervention. Palliat Med. 2011 Apr;25(3):197-209. doi: 10.1177/0269216310391691. Epub 2011 Jan 12. PMID 21228087
- [Background] Schulz R, Boerner K, Klinger J, Rosen J. Preparedness for death and adjustment to bereavement among caregivers of recently placed nursing home residents. J Palliat Med. 2015 Feb;18(2):127-33. doi: 10.1089/jpm.2014.0309. Epub 2014 Dec 3. PMID 25469737
- [Background] Schulz R, Mendelsohn AB, Haley WE, Mahoney D, Allen RS, Zhang S, Thompson L, Belle SH; Resources for Enhancing Alzheimer's Caregiver Health Investigators. End-of-life care and the effects of bereavement on family caregivers of persons with dementia. N Engl J Med. 2003 Nov 13;349(20):1936-42. doi: 10.1056/NEJMsa035373. PMID 14614169
- [Background] Steinhauser KE, Christakis NA, Clipp EC, McNeilly M, Grambow S, Parker J, Tulsky JA. Preparing for the end of life: preferences of patients, families, physicians, and other care providers. J Pain Symptom Manage. 2001 Sep;22(3):727-37. doi: 10.1016/s0885-3924(01)00334-7. PMID 11532586
- [Background] Tabachnick, B. G. and L. S. Fidell (1989). Using Multivariate Statistics, 2nd Edition. New York, Harper & Row.
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Koenig HG, Büssing A. The Duke University Religion Index (DUREL): A Five-Item Measure for Use in Epidemological Studies. Religions 1: 78-85, 2010.
- [Derived] Moore KJ, Crawley S, Fisher E, Cooper C, Vickerstaff V, Sampson EL. Exploring how family carers of a person with dementia manage pre-death grief: A mixed methods study. Int J Geriatr Psychiatry. 2023 Mar;38(3):e5867. doi: 10.1002/gps.5867. PMID 36862574
- [Derived] Moore KJ, Crawley S, Vickerstaff V, Cooper C, King M, Sampson EL. Is preparation for end of life associated with pre-death grief in caregivers of people with dementia? Int Psychogeriatr. 2020 Jun;32(6):753-763. doi: 10.1017/S1041610220000289. Epub 2020 Apr 3. PMID 32241317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11/01/2018-31/01/2019 Carers were recruited via a number of avenues including; 9 NHS hospital trusts across England who acted as Participant Identification Centres, the Join Dementia Research (JDR) website and through Alzheimer's Society avenues such as the Alzheimer's Society research network and the Care and Cure magazine.
Groups:
- All Study Participants: All Study Participants/Usual care
Period: Overall Study
Arm/Group | All Study Participants
Started | 150
Completed | 150
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White British | 131
  Ethnicity: White Other | 9
  Ethnicity: Mixed race- White and Asian | 3
  Ethnicity: Asian/Asian British - Indian | 3
  Ethnicity: Asian/Asian British - Pakistani | 1
  Ethnicity: African | 1
  Ethnicity: Declined to answer | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 150
Marital status [Count of Participants; unit: Participants]
  Single | 17
  Married/cohabitating | 124
  Divorced/separated | 8
  Widowed | 1
Relationship to person with dementia [Count of Participants; unit: Participants]
  Spouse/partner | 70
  Adult child | 72
  Other | 8
Rurality [Count of Participants; unit: Participants]
  Urban Major Conurbation | 70
  Urban City and Town | 61
  Urban City and Town in a sparse setting | 1
  Rural Town and Fringe | 9
  Rural Village | 5
  Rural Hamlets and Isolated Dwellings | 3
  Missing | 1
Deprivation [Count of Participants; unit: Participants] — Deprivation (IMD deciles) 1= most deprived 10= least deprived
  Participants
    1 | 5
    2 | 9
    3 | 9
    4 | 17
    5 | 15
    6 | 11
    7 | 15
    8 | 17
    9 | 22
    10 | 29
    Missing | 1
Employment status [Count of Participants; unit: Participants] — Question asked: Do you currently work for pay
  Participants
    Yes | 98
    No | 52
Support provided by carer [Count of Participants; unit: Participants] — Participants could select as many options were appropriate. ADL: Activities of daily living. IADL: Instrumental activities of daily living ie shopping
  Participants
    Emotional support | 147
    ADLs | 54
    IADL | 144
    Supervision | 114
Years of education [Mean (Standard Deviation); unit: years] | 16.2 (4)
Person with dementia gender [Count of Participants; unit: Participants]
  Male | 82
  Female | 68
Person with dementia age [Mean (Standard Deviation); unit: years] | 80.3 (9.7)
Does the person with dementia require constant supervision [Count of Participants; unit: Participants]
  Yes | 70
  No | 70
  Other | 9
  Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Pre-death Grief in Dementia Caregiving
Description: Marwit-Meuser Caregiver Grief Inventory Short Form (MMCGI-SF) (Marwit and Meuser 2005). 18 items with a score range from 18-90. Higher scores indicate higher levels of grief from carers of people with dementia.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 150
score on a scale | 57.6 (4.7)
Statistical Analysis 1: Comparison: All Study Participants; Test type: Other — Multivariable regression analysis will be used to enable us to explore the impact of modifiable factors reflecting preparation for end of life on the MMCGI-SF; p < 0.05, Regression, Linear; Multivariable regression will be used to explore preparation for end of life on the MMCGI-SF. The analyses will use the MMCGI-SF as the dependent variable with five predictor variables (dementia knowledge [DKAS], Social support [HLQ1], Communication with healthcare professionals [HLW4], advance decisions and knowledge of end of life wishes of person with dementia. There will also be 10 confounders included in the model (gender of caregiver, living arrangement of person with dementia [at home of a care home], aged of person with dementia, dementia severity [CDR], change in closeness, religiosity [DURAL], deprivation and relationship of the carer to the person with dementia)

2. Secondary Outcome: Knowledge of How Dementia Progresses
Description: Dementia Knowledge Assessment Scale (Annear, Toye et al. 2015). Possible score range 0-50 with a higher score indicating better knowledge of dementia.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 150
score on a scale | 34.8 (7.0)

3. Secondary Outcome: Knowledge of the Person With Dementia's End of Life Preferences
Description: Two categorical questions will be used: 'Have you had discussions with the person with dementia regarding their wishes at the end of life? (yes/no). Do you feel you have a good understanding of their wishes for end of life care? (yes/not sure/no).
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 150
Participants
  Yes | 110
  Not sure | 29
  No | 11

4. Secondary Outcome: Advance Decisions in Place for Person With Dementia
Description: Binary variable - either have or do not have any form of advance plan (such as Power of Attorney, Advance decisions to refuse treatment, Do Not attempt Resuscitation, Advance Care plan) in place for the person with dementia.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 150
Participants
  Yes | 63
  Not sure | 8
  No | 79

5. Secondary Outcome: Communication With Healthcare Providers
Description: Health Literacy Questionnaire (Osborne et al. 2013) Subscale 1 'Feeling understood and supported by healthcare providers' a Average score of 4 items leading to a range of 1-4 with higher scores indicating areas of strength.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 150
score on a scale | 2.7 (0.7)

6. Secondary Outcome: Social Support for Health Subscale of the Health Literacy Questionnaire
Description: Health Literacy Questionnaire (Osborne, Batterham et al. 2013) Sub-scale examines satisfaction with support for health from social network. Score is calculated as an average of the 5 items of the subscale leading to a score range of 1-4 with higher scores indicating that a person's social system provides them with all the support they want or need.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 150
score on a scale | 2.7 (0.6)

7. Secondary Outcome: Dementia Severity
Description: Carer report of their relative/friend's severity of dementia using the Clinical Dementia Rating scale (Morris 1993). This scale leads to scores 5 possible scores; 0=no dementia, 0.5=questionable dementia, 1=mild dementia, 2=moderate dementia and 3=severe dementia.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 150
Participants
  Questionable dementia | 4
  Mild dementia | 34
  Moderate dementia | 64
  Severe dementia | 48

8. Secondary Outcome: Intrinsic Religiosity
Description: Duke University Religion Index (Koenig and Büssing 2010). Using the subscale 'Intrinsic religiosity' which assesses degree of personal religious commitment or motivation which has been more strongly associated with protecting from psychological distress. Possible score range is 0-12 with a higher score indicating a stronger personal religious commitment/motivation.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 150
score on a scale | 6.6 (4.3)

ADVERSE EVENTS:
Time Frame: One interview
Groups:
- All Study Participants: All Study Participants/ Usual care
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/150
Serious Adverse Events (participants affected / at risk) | 0/150
Other Adverse Events (participants affected / at risk) | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT03332979/Prot_SAP_000.pdf